CLINICAL TRIAL: NCT00877552
Title: Prospective Studies of the Pathogenesis of Schizophrenia (Center Title) Early Brain Development in High Risk Children (Project Title) Early Brain Development in One and Two Year Olds (Associated Grant Title)
Brief Title: Prospective Studies of the Pathogenesis of Schizophrenia
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 04-1144; R01HD053000-02 (NIH); P50MH064065-07 (NIH)
Record Dates: First submitted 2009-04-06; First posted 2009-04-08 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; brain development; MRI
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — MRIs, buccal swabs, prenatal ultrasounds
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control: Typically developing
- Mild ventriculomegaly (MVM): Fetal isolated mild ventriculomegaly
- Schizophrenia High Risk: Offspring of mothers with schizophrenia
- Bipolar High Risk: Offspring of mothers with schizophrenia

SUMMARY:
The purpose of this study is to use structural and functional magnetic resonance imaging (MRI) to study children at high risk for schizophrenia. It is hypothesized that children at high risk for schizophrenia will have abnormalities of brain development, especially of the cerebral cortex. The study will also describe normal brain development in children from birth to age 6 years

DETAILED DESCRIPTION:
We are currently following enrolled children at 4 and 6 years of age. We are obtaining structural MRIs and rsfMRIs. In addition, we are assessing cognitive function and behavior with Stanford-Binet, BRIEF and BASC.

ELIGIBILITY:
Inclusion Criteria:

* control, offspring of mother with schizophrenia or bipolar illness; child with MVM

Exclusion Criteria:

* major neurological or medical illness

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: medical center and community clinics
Sampling Method: Non-Probability Sample
Enrollment: 598 (Actual)
Dates: Start 2002-08; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
magnetic resonance images (structural and functional) | birth, ages 1, 2 , 4 and 6 years

SECONDARY OUTCOMES:
Cognitive development | 0,1,2,4 and 6 years

CONTACTS AND LOCATIONS:
Overall Officials: John Gilmore, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Department of Psychiatry, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Gilmore JH. Understanding what causes schizophrenia: a developmental perspective. Am J Psychiatry. 2010 Jan;167(1):8-10. doi: 10.1176/appi.ajp.2009.09111588. No abstract available. PMID 20068120
- [Background] Alcauter S, Lin W, Smith JK, Short SJ, Goldman BD, Reznick JS, Gilmore JH, Gao W. Development of thalamocortical connectivity during infancy and its cognitive correlations. J Neurosci. 2014 Jul 2;34(27):9067-75. doi: 10.1523/JNEUROSCI.0796-14.2014. PMID 24990927
- [Background] Knickmeyer RC, Meltzer-Brody S, Woolson S, Hamer RM, Smith JK, Lury K, Gilmore JH. Rate of Chiari I malformation in children of mothers with depression with and without prenatal SSRI exposure. Neuropsychopharmacology. 2014 Oct;39(11):2611-21. doi: 10.1038/npp.2014.114. Epub 2014 May 20. PMID 24837031
- [Background] Li G, Wang L, Shi F, Lyall AE, Lin W, Gilmore JH, Shen D. Mapping longitudinal development of local cortical gyrification in infants from birth to 2 years of age. J Neurosci. 2014 Mar 19;34(12):4228-38. doi: 10.1523/JNEUROSCI.3976-13.2014. PMID 24647943
- [Background] Girault JB, Cornea E, Goldman BD, Knickmeyer RC, Styner M, Gilmore JH. White matter microstructural development and cognitive ability in the first 2 years of life. Hum Brain Mapp. 2019 Mar;40(4):1195-1210. doi: 10.1002/hbm.24439. Epub 2018 Oct 24. PMID 30353962
- [Background] Girault JB, Langworthy BW, Goldman BD, Stephens RL, Cornea E, Reznick JS, Fine J, Gilmore JH. The Predictive Value of Developmental Assessments at 1 and 2 for Intelligence Quotients at 6. Intelligence. 2018 May-Jun;68:58-65. doi: 10.1016/j.intell.2018.03.003. Epub 2018 Mar 16. PMID 30270948
- [Background] Knickmeyer RC, Xia K, Lu Z, Ahn M, Jha SC, Zou F, Zhu H, Styner M, Gilmore JH. Impact of Demographic and Obstetric Factors on Infant Brain Volumes: A Population Neuroscience Study. Cereb Cortex. 2017 Dec 1;27(12):5616-5625. doi: 10.1093/cercor/bhw331. PMID 27797836
- [Result] Knickmeyer RC, Gouttard S, Kang C, Evans D, Wilber K, Smith JK, Hamer RM, Lin W, Gerig G, Gilmore JH. A structural MRI study of human brain development from birth to 2 years. J Neurosci. 2008 Nov 19;28(47):12176-82. doi: 10.1523/JNEUROSCI.3479-08.2008. PMID 19020011
- [Result] Gao W, Lin W, Chen Y, Gerig G, Smith JK, Jewells V, Gilmore JH. Temporal and spatial development of axonal maturation and myelination of white matter in the developing brain. AJNR Am J Neuroradiol. 2009 Feb;30(2):290-6. doi: 10.3174/ajnr.A1363. Epub 2008 Nov 11. PMID 19001533
- [Result] Gilmore JH, Smith LC, Wolfe HM, Hertzberg BS, Smith JK, Chescheir NC, Evans DD, Kang C, Hamer RM, Lin W, Gerig G. Prenatal mild ventriculomegaly predicts abnormal development of the neonatal brain. Biol Psychiatry. 2008 Dec 15;64(12):1069-76. doi: 10.1016/j.biopsych.2008.07.031. Epub 2008 Oct 2. PMID 18835482
- [Result] Gilmore JH, Lin W, Corouge I, Vetsa YS, Smith JK, Kang C, Gu H, Hamer RM, Lieberman JA, Gerig G. Early postnatal development of corpus callosum and corticospinal white matter assessed with quantitative tractography. AJNR Am J Neuroradiol. 2007 Oct;28(9):1789-95. doi: 10.3174/ajnr.a0751. PMID 17923457
- [Result] Lin W, Zhu Q, Gao W, Chen Y, Toh CH, Styner M, Gerig G, Smith JK, Biswal B, Gilmore JH. Functional connectivity MR imaging reveals cortical functional connectivity in the developing brain. AJNR Am J Neuroradiol. 2008 Nov;29(10):1883-9. doi: 10.3174/ajnr.A1256. Epub 2008 Sep 10. PMID 18784212
- [Result] Gilmore JH, Lin W, Prastawa MW, Looney CB, Vetsa YS, Knickmeyer RC, Evans DD, Smith JK, Hamer RM, Lieberman JA, Gerig G. Regional gray matter growth, sexual dimorphism, and cerebral asymmetry in the neonatal brain. J Neurosci. 2007 Feb 7;27(6):1255-60. doi: 10.1523/jneurosci.3339-06.2007. PMID 17287499
- [Result] Looney CB, Smith JK, Merck LH, Wolfe HM, Chescheir NC, Hamer RM, Gilmore JH. Intracranial hemorrhage in asymptomatic neonates: prevalence on MR images and relationship to obstetric and neonatal risk factors. Radiology. 2007 Feb;242(2):535-41. doi: 10.1148/radiol.2422060133. Epub 2006 Dec 19. PMID 17179400
- [Result] Gilmore JH, Kang C, Evans DD, Wolfe HM, Smith JK, Lieberman JA, Lin W, Hamer RM, Styner M, Gerig G. Prenatal and neonatal brain structure and white matter maturation in children at high risk for schizophrenia. Am J Psychiatry. 2010 Sep;167(9):1083-91. doi: 10.1176/appi.ajp.2010.09101492. Epub 2010 Jun 1. PMID 20516153
- [Result] Shi F, Yap PT, Wu G, Jia H, Gilmore JH, Lin W, Shen D. Infant brain atlases from neonates to 1- and 2-year-olds. PLoS One. 2011 Apr 14;6(4):e18746. doi: 10.1371/journal.pone.0018746. PMID 21533194
- [Result] Gao W, Zhu H, Giovanello KS, Smith JK, Shen D, Gilmore JH, Lin W. Evidence on the emergence of the brain's default network from 2-week-old to 2-year-old healthy pediatric subjects. Proc Natl Acad Sci U S A. 2009 Apr 21;106(16):6790-5. doi: 10.1073/pnas.0811221106. Epub 2009 Apr 7. PMID 19351894
- [Result] Short SJ, Elison JT, Goldman BD, Styner M, Gu H, Connelly M, Maltbie E, Woolson S, Lin W, Gerig G, Reznick JS, Gilmore JH. Associations between white matter microstructure and infants' working memory. Neuroimage. 2013 Jan 1;64:156-66. doi: 10.1016/j.neuroimage.2012.09.021. Epub 2012 Sep 16. PMID 22989623
- [Result] Geng X, Gouttard S, Sharma A, Gu H, Styner M, Lin W, Gerig G, Gilmore JH. Quantitative tract-based white matter development from birth to age 2years. Neuroimage. 2012 Jul 2;61(3):542-57. doi: 10.1016/j.neuroimage.2012.03.057. Epub 2012 Mar 28. PMID 22510254
- [Result] Gilmore JH, Shi F, Woolson SL, Knickmeyer RC, Short SJ, Lin W, Zhu H, Hamer RM, Styner M, Shen D. Longitudinal development of cortical and subcortical gray matter from birth to 2 years. Cereb Cortex. 2012 Nov;22(11):2478-85. doi: 10.1093/cercor/bhr327. Epub 2011 Nov 22. PMID 22109543
- [Result] Lyall AE, Woolson S, Wolfe HM, Goldman BD, Reznick JS, Hamer RM, Lin W, Styner M, Gerig G, Gilmore JH. Prenatal isolated mild ventriculomegaly is associated with persistent ventricle enlargement at ages 1 and 2. Early Hum Dev. 2012 Aug;88(8):691-8. doi: 10.1016/j.earlhumdev.2012.02.003. Epub 2012 Mar 22. PMID 22445211
- [Result] Lyall AE, Shi F, Geng X, Woolson S, Li G, Wang L, Hamer RM, Shen D, Gilmore JH. Dynamic Development of Regional Cortical Thickness and Surface Area in Early Childhood. Cereb Cortex. 2015 Aug;25(8):2204-12. doi: 10.1093/cercor/bhu027. Epub 2014 Mar 2. PMID 24591525
- [Result] Knickmeyer RC, Wang J, Zhu H, Geng X, Woolson S, Hamer RM, Konneker T, Lin W, Styner M, Gilmore JH. Common variants in psychiatric risk genes predict brain structure at birth. Cereb Cortex. 2014 May;24(5):1230-46. doi: 10.1093/cercor/bhs401. Epub 2013 Jan 2. PMID 23283688